CLINICAL TRIAL: NCT00956215
Title: A Randomized and Placebo-Controlled Evaluation of Aprepitant for Decreasing the Incidence of Post-Operative Nausea and Vomiting (PONV) in Bariatric Patients
Brief Title: Decreasing the Incidence of Post-Operative Nausea and Vomiting (PONV) in Bariatric Patients
Acronym: PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Emend
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Nausea; Vomiting
Keywords: post operative; obese
MeSH Terms: conditions — Nausea; Vomiting; Obesity | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 80mg of Aprepitant (Active Comparator): Patients will be randomized to receive 80mg of Aprepitant with 50 ml of water no later than 30 minutes before induction of anesthesia.
  Interventions: Drug: Aprepitant
- 80 mg of placebo (Placebo Comparator): . Patients will be randomized to placebo with 50 ml of water no later than 30 minutes before induction of anesthesia.
  Interventions: Drug: Aprepitant placebo

INTERVENTIONS:
Drug: Aprepitant — 80 mg tablet of Aprepitant with 50 ml of water 30 minutes before surgery
  Arms: 80mg of Aprepitant
Drug: Aprepitant placebo — 80 mg placebo tablet with 50 ml of water no later than 30 minutes before induction of anesthesia.
  Arms: 80 mg of placebo

SUMMARY:
The study drug, Aprepitant, is currently used to control chemotherapy induced nausea and vomiting and is also approved for post-operative nausea and vomiting. The investigators' evaluation of it in morbidly obese patients will demonstrate its ability to control nausea and vomiting post-operatively in this subset of patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of Aprepitant, also known as Emend, in reducing post-operative nausea and vomiting in morbidly obese patients. Post-operative nausea and vomiting that occurs in morbidly obese patients can greatly increase the chances of complications during the post-operative period. By treating morbidly obese patients with Aprepitant, the goal is to reduce the risk of such complications that may be induced by nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

Subjects included in this study must be:

* Female
* At least 18 years of age
* Non-smoking
* At high risk for PONV
* Obese with a BMI of at least 45 kg/m2
* Undergoing upper gastrointestinal surgery requiring postoperative opioid analgesia

Exclusion Criteria:

Subjects will be excluded if:

* They have a known allergy to Aprepitant or Ondansetron
* They are currently taking Orap (pimozide), Seldane (terfenadine), Hismanal (astemizole), or Propulsid (cisapride)
* They are pregnant
* They are breastfeeding
* They plan on getting pregnant in the 2 months following surgery
* They are not able to receive patient controlled analgesia (PCA) following surgery
* They have a known drug or alcohol abuse problem
* They have chronic nausea and vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of 80mg Aprepitant in preventing post operative nausea or vomiting in morbidly obese patients (BMI of 45 kg/m2 or higher) undergoing upper gastrointestinal surgery. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Sinha, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States